CLINICAL TRIAL: NCT03201757
Title: A Phase 3 Study to Assess the Long Term Safety, Tolerability, and Durability of Treatment Effect of ALKS 3831 in Subjects With Schizophrenia, Schizophreniform Disorder, or Bipolar I Disorder
Brief Title: Study to Evaluate the Long-term Safety, Tolerability, and Durability of Treatment Effect of ALKS 3831
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALK3831-A308
Record Dates: First submitted 2017-06-15; First posted 2017-06-28 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-08

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Bipolar I Disorder
Keywords: Alkermes; ALKS 3831; Olanzapine; Samidorphan; Schizophrenia; Schizophreniform; Bipolar I
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALKS 3831 (Experimental): Coated bilayer tablet
  Interventions: Drug: ALKS 3831

INTERVENTIONS:
Drug: ALKS 3831 — Olanzapine + samidorphan, daily oral dosing

SUMMARY:
This study will evaluate the long-term safety, tolerability, and durability of treatment effect of ALKS 3831 in subjects with schizophrenia, schizophreniform disorder, or bipolar I disorder

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent/assent as per local requirements
* Agrees to use an acceptable method of contraception during the study, and for 30 days after any study drug administration, unless surgically sterile or post-menopausal
* Has the potential to benefit from the administration of ALKS 3831, in the opinion of the investigator
* Subject met the eligibility criteria of the antecedent study at the time of enrollment in the antecedent study and completed the treatment period in one of the following antecedent studies within 7 days: ALK3831-A304, ALK3831-A306, or ALK3831-A307
* Additional criteria may apply

Exclusion Criteria:

* Has any finding that, in the view of the investigator or medical monitor, would compromise the safety of the subject or affect their ability to fulfill the protocol visit schedule or visit requirements
* Has a positive drug screen for drugs of abuse at study entry
* Currently pregnant or breastfeeding or is planning to become pregnant during the study or within 30 days of the last study drug administration
* Additional criteria may apply

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (79):
- United States (43):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Rogers, Arkansas
  - Alkermes Investigational Site, Anaheim, California
  - Alkermes Investigational Site, Cerritos, California
  - Alkermes Investigational Site, Culver City, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, Glendale, California
  - Alkermes Investigational Site, Long Beach, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Palo Alto, California
  - Alkermes Investigational Site, Pico Rivera, California
  - Alkermes Investigational Site, Redlands, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Temecula, California
  - Alkermes Investigational Site, Torrance, California
  - Alkermes Investigational Site, Lauderhill, Florida
  - Alkermes Investigational Site, North Miami, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Augusta, Georgia
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Winfield, Illinois
  - Alkermes Investigational Site, Grand Rapids, Michigan
  - Alkermes Investigational Site, Flowood, Mississippi
  - Alkermes Investigational Site, Kansas City, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Berlin, New Jersey
  - Alkermes Investigational Site, Marlton, New Jersey
  - Alkermes Investigational Site, Brooklyn, New York
  - Alkermes Investigational Site, Rochester, New York
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Cincinnati, Ohio
  - Alkermes Investigational Site, Dayton, Ohio
  - Alkermes Investigational Site, Eugene, Oregon
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Fort Worth, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Richardson, Texas
  - Alkermes Investigational Site, Bellevue, Washington
- Alkermes Investigational Site, Vienna, Austria
- Bulgaria (8):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Lovech
  - Alkermes Investigational Site, Novi Iskar
  - Alkermes Investigational Site, Plovdiv
  - Alkermes Investigational Site, Sofia
  - Alkermes Investigational Site, Tserova Koria
  - Alkermes Investigational Site, Veliko Tarnovo
  - Alkermes Investigational Site, Vratsa
- Alkermes Investigational Site, Galway, Ireland
- Israel (2):
  - Alkermes Investigational Site, Jerusalem
  - Alkermes Investigational Site, Ramat Gan
- Italy (2):
  - Alkermes Investigational Site, Brescia
  - Alkermes Investigational Site, Napoli
- Alkermes Investigational Site, Poznan, Poland
- Alkermes Investigational Site, San Juan, Puerto Rico
- Russia (8):
  - Alkermes Investigational Site, Arkhangelsk
  - Alkermes Investigational Site, Moscow
  - Alkermes Investigational Site, Roshchino
  - Alkermes Investigational Site, Rostov-on-Don
  - Alkermes Investigational Site, Saint Petersburg
  - Alkermes Investigational Site, Samara
  - Alkermes Investigational Site, Saratov
  - Alkermes Investigational Site, Tonnel’nyy
- Serbia (3):
  - Alkermes Investigational Site, Belgrade
  - Alkermes Investigational Site, Kragujevac
  - Alkermes Investigational Site, Novi Kneževac
- Alkermes Investigational Site, Busan, South Korea
- Ukraine (7):
  - Alkermes Investigational Site, Kharkiv
  - Alkermes Investigational Site, Kherson
  - Alkermes Investigational Site, Kyiv
  - Alkermes Investigational Site, Lviv
  - Alkermes Investigational Site, Poltava
  - Alkermes Investigational Site, Smila
  - Alkermes Investigational Site, Vinnytsia
- Alkermes Investigational Site, Headington, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ballon JS, Kahn RS, Arevalo C, Dunbar M, McDonnell D, Correll CU. Long-Term Safety, Tolerability, and Durability of Treatment Effect of Olanzapine and Samidorphan: Results of a 4-Year Open-Label Study. J Clin Psychiatry. 2024 Dec 4;86(1):24m15511. doi: 10.4088/JCP.24m15511. PMID 39630083

RESULTS

PARTICIPANT FLOW:
Groups:
- ALKS 3831: Coated bilayer tablet
  ALKS 3831: Olanzapine + samidorphan, daily oral dosing ranging from 5/10, 10/10, 15/10, and 20/10 mg at the Investigator's discretion.
Period: Overall Study
Arm/Group | ALKS 3831
Started | 523
Completed | 188
Not Completed | 335
Not completed — Withdrawal by Subject | 133
Not completed — Adverse Event | 44
Not completed — Lost to Follow-up | 37
Not completed — Pregnancy | 2
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 20
Not completed — Study Terminated at Site by Sponsor Due to Regional War | 1
Not completed — Not Yet Determined | 5
Not completed — Logistical Difficulties Due to Regional Wars & COVID-19 | 72
Not completed — Other | 20

BASELINE CHARACTERISTICS:
Population: All analyses were conducted using the safety population except for the analyses of adverse events in the safety follow up period
Arm/Group | ALKS 3831
Number analyzed (Participants) | 523
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201
  Male | 322
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 504
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 126
  White | 380
  More than one race | 7
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 206
  Ukraine | 118
  United Kingdom | 2
  Russia | 69
  Austria | 2
  South Korea | 2
  Ireland | 2
  Poland | 2
  Italy | 4
  Israel | 28
  Bulgaria | 63
  Serbia | 25
Height [Mean (Standard Deviation); unit: Centimeters] | 172.28 (9.481)
Weight [Mean (Standard Deviation); unit: kilograms] | 77.39 (15.486)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.00 (4.332)
Clinical Global Impression-Severity [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression (CGI) is a 3-item, clinician-rated scale used to assess global illness severity, overall improvement from the start of treatment, and therapeutic response. Rate a participant 1-7; from "not at all ill" (ie, score of 1) to "among the most extremely ill" (ie, score of 7)
  units on a scale | 3.06 (.867)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Time Frame: Up to 48 months
Population: All enrolled participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 3831
Number analyzed (Participants) | 523
Participants | 314

2. Primary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Scale
Description: The clinical global impression - severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis; 1 being normal, not ill at all and 7 being among the severally ill patients
Time Frame: Up to 48 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ALKS 3831
Number analyzed (Participants) | 523
units on a scale | -.24 (.651)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the treatment period (24- 48 months) and through-out the safety follow-up period (4 weeks);
Arm/Group | ALKS 3831
All-Cause Mortality (participants affected / at risk) | 1/523
Serious Adverse Events (participants affected / at risk) | 35/523
Other Adverse Events (participants affected / at risk) | 314/523
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ALKS 3831 (N=523)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Infected naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Drug withdrawal convulsions (Nervous system disorders) | 1 (1)
Intracranial aneursym (Nervous system disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 11 (11)
Anxiety (Psychiatric disorders) | 2 (2)
Acute psychosis (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1)
Depression Suicidal (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Psychiatric symptom (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Psychotic symptom (Psychiatric disorders) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALKS 3831 (N=523)
Weight increased (Investigations) | 51
Headache (Nervous system disorders) | 37
Anxiety (Psychiatric disorders) | 32
Insomnia (Psychiatric disorders) | 31
Nausea (Gastrointestinal disorders) | 30
Weight decreased (Investigations) | 30
Blood creatine phosphokinase increased (Investigations) | 22
Nasopharyngitis (Infections and infestations) | 17
Schizophrenia (Psychiatric disorders) | 15
Vomiting (Gastrointestinal disorders) | 15
Blood triglycerides increased (Investigations) | 14
Constipation (Gastrointestinal disorders) | 13
Low density lipoprotein increased (Investigations) | 13
Upper respiratory tract infection (Infections and infestations) | 13
Alanine aminotransferase increased (Investigations) | 12
Blood prolactin increased (Investigations) | 12
Dizziness (Nervous system disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT03201757/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT03201757/SAP_001.pdf